CLINICAL TRIAL: NCT00559728
Title: Magnetic Resonance Imaging (MRI) Analysis of Coronary Artery Plaque Components
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_3763
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Artery Plaque Components

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze atherosclerotic vessel wall components with multidetector computed tomography (MDCT) and compare with MRI. The hypothesis is that MRI is comparable to computed tomography (CT) in showing plaque components of coronary plaques.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females 18 - 65 who are scheduled to undergo a CT scan for evaluation of coronary artery plaque.

Exclusion Criteria:

* Contraindications to having an MRI scan
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Females 18 - 65 scheduled to undergo a clinically-indicated coronary artery CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Bluemke, MD, PhD, Principal Investigator — Johns Hopkins University